CLINICAL TRIAL: NCT03918694
Title: Vitamin C Supplementation for Lumbar Spine Surgical Patients
Brief Title: Vitamin C Supplement for Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00143319
Record Dates: First submitted 2019-01-04; First posted 2019-04-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spine Surgery
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: 2 groups: placebo and Vitamin C
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Blinded pilot randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): Participants will receive Vit C tablets
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Participants will receive placebo tablets
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Daily use of Vit C tablets
  Arms: Experimental
Dietary Supplement: Placebo — Daily use of placebo tablets
  Arms: Placebo

SUMMARY:
By doing this study, researchers hope to learn effects of Vit C on lumbar spine surgery outcomes.

DETAILED DESCRIPTION:
Lumbar spine surgeries are common procedures for management of low back pain and their prevalence is increasing. However, their outcomes are less than optimal.

An effective and inexpensive solution to minimizing surgical complications and expediting recovery following lumbar spine surgery could be supplementation using high doses of vitamin C, also known as ascorbic acid. Vit C can help reduce oxidative stress and inflammation and improve immune system and body's own chemicals to fight pain.

The researchers want to examine if Vit C is effective in decreasing pain and pain medications and improving function. Gaining a better understanding of effects of Vit C on patient recovery may lead to improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to have a lumbar spine fusion
* Can read and understand the English language
* BMI 35 or less

Exclusion Criteria:

* Patients taking certain medications
* lumbar spine laminectomy or discectomy
* taking a Vit C supplement
* pregnancy
* Cauda equine syndrome or spinal tumor
* neurological, neurodegenerative or cognitive issues
* renal pathology
* sickle cell anemia
* iron metabolism disorder

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility outcome | up to 7 weeks
  The number of participants recruited and enrolled.
Adherence feasibility outcome | up to 7 weeks
  Calculate adherence in percentage as subjects enrolled versus completed
Pain intensity: numeric rating pain scale | up to 7 weeks
  self reported 0-10 numeric rating pain scale where 0=no pain and 10=most pain imagined
Pain medication consumption | up to 7 weeks
  Use of opioids and non-opioids analgesics documented in patients' health records
Function | up to 7 weeks
  Gait distance in feet will be obtained during physical therapy visit
Would healing | up to 7 weeks
  Surgical incision observation

SECONDARY OUTCOMES:
Beck depression inventory | up to 7 weeks
  A standard questionnaire with 1 - 40 points, 1=no depression and 40=extreme depression
Vit C level | up to 7 weeks
  Serum level of Vit C in umol/L
Beck anxiety inventory | up to 7 weeks
  A standard questionnaire with 21 questions. Scores 0-21=low anxiety, scores 22-35=moderate anxiety and scores 36 and above=potentially concerning level of anxiety
2011 Fibromyalgia (FM) survey | up to 7 weeks
  A standard questionnaire for centralized pain. Scores 3-6 in widespread pain index and 9 or greater in symptom severity suggest widespread pain
fatigue questionnaire | up to 7 weeks
  A standard questionnaire with 10 fatigue related questions. Each measured on 1-5 Likert scale. Higher numbers indicate greater fatigue
Pittsburg sleep scale | up to 7 weeks
  A standard questionnaires to examine sleep problems. A total of 5 scores or greater indicate poor sleep quality
Pain catastrophizing scale | up to 7 weeks
  A standard scale to measure catastrophizing thoughts. Higher numbers indicate greater catastrophizing thoughts

CONTACTS AND LOCATIONS:
Overall Officials: Neena Sharma, PT, PhD, CMPT, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No